CLINICAL TRIAL: NCT00213863
Title: Implantation of Porous Titanium Prosthesis in Laryngeal Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3097
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Vocal Cord Paralysis
Keywords: porous titanium implants; thyroplasty; vocal cord paralysis; male or female more than 18 years old
MeSH Terms: conditions — Vocal Cord Paralysis | interventions — Laryngoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vocal fold medialization (thyroplasty) prosthesis by insertion of a new implant allowing very easy and quick setting — The porous titanium prosthesis is implanted under local anaesthesia. Neck incision is performed in order to expose the thyroidal cartilage. A window is then opened in this cartilage, and the implant is placed in contact with the vocal muscles. The patient is then asked to speak in order to achieve the implant best setting.

SUMMARY:
This study evaluates a medialization implant to treat vocal cord paralysis, to permit it to adjust the quality of the voice under local or general anesthesia. The aim is to restore phonation using a porous titanium prosthesis in laryngeal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than 18 years old

Exclusion Criteria:

* Age less than 18 years
* Pregnant women
* Local carcinoma excluding radiotherapeutic or surgical control
* Bad general condition
* Contraindication to general anesthesia
* Non-controlled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Nasofibroscopy | 8 days and 3 months after surgery
Voice control and recording | 8, 15, 30 days, 3, 6 months after surgery and then, every 6 months during the whole trial
All types of complication | 8, 15, 30 days, 3, 6 months after surgery and then, every 6 months during the whole trial

CONTACTS AND LOCATIONS:
Overall Officials: Christian Debry, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (1):
- Service d'Oto-Rhino-Laryngologie et de Chirurgie Cervico-Faciale, Hôpital de Hautepierre, Strasbourg, France